CLINICAL TRIAL: NCT02418468
Title: Effects of Indacaterol in Symptomatic COPD Patients With Low Risk of Exacerbations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149BHK02
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, FEV1, indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): Matching placebo indacaterol capsules for inhalation once daily delivered via the Novartis single dose dry power inhaler (SDDPI) (Onbrez® Breezhaler®)
  Interventions: Drug: Placebo
- Indacaterol 150 mcg (Experimental): Indacaterol 150 mcg capsules for inhalation once daily delivered via the Novartis single dose dry power inhaler (SDDPI) (Onbrez® Breezhaler®)
  Interventions: Drug: Indacaterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150µg capsules for inhalation daily
  Arms: Indacaterol 150 mcg
Drug: Placebo — Matching placebo indacaterol capsules for inhalation daily
  Arms: Placebo

SUMMARY:
This study compared the efficacy of indacaterol versus placebo in COPD patients classified as GOLD 2014 Patient Group B.

This was a 2-arm parallel group study that recruited COPD patients classified by GOLD Patient Gorup B. On successful completion of run-in period, patients were randomized in the ratio 1:1 to receive prn salbutamol plus:

1. Indacaterol 150ug or
2. Placebo for indacaterol all once daily (od) for 26 weeks. The primary objective (trough FEV1) was assessed after 12 weeks.

ELIGIBILITY:
Inclusion criteria

1. Male or female adults aged ≥40 years, who have provided their consent and signed an Informed Consent Form. Written informed consent must be obtained before any assessment is performed.
2. Patients diagnosed with COPD at 40 years of age or older.
3. Patients with smoking history of at least 10 pack years, both current and ex-smokers are eligible. (Ten pack years is defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years, etc)
4. Patients with stable COPD in Patient Group B according to GOLD 2014.

Exclusion criteria

1. Use of other investigational drugs within 5 half-lives of enrollment, or [within 30 days /until the expected PD effect has returned to baseline], whichever is longer.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
4. Patients who have had 2 or more COPD exacerbations that required treatment with antibiotics, systemic steroids (oral or intravenous) or 1 or more exacerbation resulting in hospitalization in the 12 months prior to Visit 1.
5. Patients who have COPD exacerbation or infection 6 weeks prior to Visit 1.
6. Patients who develop a moderate or severe COPD exacerbation during the period between Visit 1 and Visit 2.
7. Patients with a history of asthma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-04-19 (Actual); Study Completion 2016-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 150 mcg | Placebo
Started | 13 | 11
Completed | 11 | 10
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal of informed consent | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 mcg | Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7.2) | 68.8 (14.96) | 66 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at 12 Weeks
Description: To compare the effects of indacaterol 150ug once dialy (od) to placebo in GOLD 2014 Group B COPD patients, in terms of 24-hour postdose (trough) forced expiratory volume in 1 second (FEV1) after 12 weeks of dosing.
Time Frame: at week 12
Population: Full Analysis Set (FAS) - would include all randomized patients who received at least one dose of study drug. Following the intent-to-treat principle, patients would be analyzed according to the treatment assigned at randomization.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 mcg | Placebo
Number analyzed (Participants) | 13 | 11
Liters | 1.76 (0.067) | 1.86 (0.061)
Statistical Analysis 1: Comparison: Indacaterol 150 mcg vs Placebo; Test type: Superiority or Other; p = 0.262, mixed models for repeated measures (MMRM; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.26 to 0.07], Standard Error of Mean 0.08

ADVERSE EVENTS:
Arm/Group | Indacaterol 150 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/13
Other Adverse Events (participants affected / at risk) | 2/11 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 mcg (N=11) | Placebo (N=13)
Influenza viral infections (Infections and infestations) | 0 | 1
Thoracic cage fractures non-spinal (Injury, poisoning and procedural complications) | 0 | 1
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 mcg (N=11) | Placebo (N=13)
Inner ear signs and sympotoms (Ear and labyrinth disorders) | 1 | 0
Corneal injuries (Eye disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorders sign and symptoms NEC (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.